CLINICAL TRIAL: NCT02067286
Title: Multi-Center Study of In Vitro Diagnostic Devices for the Detection of Influenza A, Influenza B, and RSV
Brief Title: Detection of Influenza A, Influenza B, and RSV Using the Liat™ Assays on the Liat™ Analyzer
Status: Completed | Type: Observational
Sponsor: IQuum, Inc. (Industry)
Collaborators: Roche Molecular Systems, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: FR4, Rev. 3.3
Record Dates: First submitted 2014-02-14; First posted 2014-02-20 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Influenza A; Influenza B; Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the clinical sensitivity and specificity of the Liat™ Influenza A/B & RSV Assay and the Liat™ Influenza A/B Assay when used on the Liat Analyzer to detect the presence or absence of Influenza A, Influenza B, and RSV in a nasopharyngeal swab specimen as compared to an FDA approved NAAT and culture.

ELIGIBILITY:
Inclusion Criteria:

* Patients exhibiting 2 or more symptom groups characteristic of influenza and/or RSV at the time of visit or within the past 48 hours:

  1. fever of at least 37.8 C (100F)
  2. runny or stuffy nose
  3. coughing, wheezing or difficulty breathing
  4. sore throat, headache, extreme tiredness, or muscle aches
  5. infants: decreased activity, irritability, poor feeding
* Subject who are able to understand and consent to participation; for minors under the age of 18, this includes a parent or legal guardian

Exclusion Criteria:

* Patients who are under-going anti-viral medication now or within the last 7 days.
* Patients who received Nasal Spray Flu Vaccine within the last 6 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must be exhibiting symptoms characteristic of influenza or RSV
Sampling Method: Non-Probability Sample
Enrollment: 1642 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the Liat™ Influenza A/B & RSV Assay and the Liat™ Influenza A/B Assay as compared to an FDA-cleared nucleic acid amplification test | 1 day

SECONDARY OUTCOMES:
Evaluate the sensitivity and specificity of the Liat™ Influenza A/B & RSV Assay and the Liat™ Influenza A/B Assay as compared to culture | 1 day

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Pediatrics-by-the-Sea, Delray Beach, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Meridian Clinical Research, Bellevue, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - Accurate Clinical Research, Houston, Texas
  - Plano Pediatrics, Plano, Texas
  - Advanced Pediatrics, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: No